CLINICAL TRIAL: NCT01785914
Title: Retrospective Evaluation of the Clinical Results Obtained in Patients With Acute Lymphoblastic Leukemia Treated at the San Giovanni Battista Hospital.
Acronym: ALL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Principal Investigator, Benedetto Bruno, MD, Azienda Ospedaliera San Giovanni Battista
Other Study IDs: ALL-TO-2012
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Disease: Acute Lymphoblastic Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This study provides for the collection of a series composed by patients with newly diagnosed of acute lymphoblastic leukemia in the period 1999-2011. This collection is carried out with retrospective investigation, through the review of paper and electronic records and data cards in large part already collected as part of study protocols "GIMEMA" or "BFM" or "NILG" approved by the Ethics Committee of Hospital. The purpose of data collection is to check with retrospective predictability of classical risk factors in relation to disease response, and overall survival of the event-free survival, to estimate the cumulative incidence of competitive events such as the emergence of disease, acute and chronic transplant, the transplant-related mortality and relapse of disease.

ELIGIBILITY:
Patients with newly diagnosed of acute lymphoblastic leukemia enrolled from 1999 to 2011 at the Division of Hematology, Molinette University Hospital and candidates for therapeutic approach with curative intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute lymphoblastic leukemia patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
Event-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Bruno, MD, Principal Investigator — Divisione di Ematologia-Città della Salute e della Scienza di Torino
Locations (1):
- Città della Salute e della Scienza di Torino, Torino, Italy